CLINICAL TRIAL: NCT02686554
Title: Elucidating the Proteostatis Network to Control Alzheimer's Disease - Identification of Proteostasis-related Biomarkers in Alzheimer´s Dementia
Brief Title: Identification of Proteostasis-related Biomarkers in Alzheimer´s Dementia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Oliver Peters, MD, MD, senior resident, Charite University, Berlin, Germany
Other Study IDs: BIH_CRG2a_TP5
Record Dates: First submitted 2016-02-16; First posted 2016-02-19 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Alzheimer Disease
Keywords: Biomarker
MeSH Terms: conditions — Alzheimer Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, cerebrospinal fluid, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AD patients
  Interventions: Other: Neuropsychological assessment
- AD patients immunized
  Interventions: Other: Neuropsychological assessment

INTERVENTIONS:
Other: Neuropsychological assessment — The patients perform tests to assess their cognitive abilities

SUMMARY:
At the time of biomarker-substantiated diagnosis for a given AD patient it remains unclear to what extent the disease will devastate cognitive abilities within the next years. This is not only unsatisfying for the patient and the attending physician but also a major problem in the context of clinical trials that aim to establish new therapeutic agents. In clinical trials it is critically important to foresee as precisely as possible the course of the disease. The overall aim of the subproject is to identify a panel of CSF biomarkers to further improve specificity of diagnosis ("disease markers"), to measure disease activity and to predict AD progression ("stage and progression markers").

DETAILED DESCRIPTION:
Within the last years, protein analyses of Aβ-species in the cerebrospinal fluid (CSF) and amyloid-imaging using F18-based PET-tracers have become a part of the diagnostic repertoire in specialized memory clinics allowing a neurobiological, biomarker-based validation of Alzheimer´s disease (AD) diagnosis. This has led to a substantial increase in the specificity of the diagnostic procedure. However, the problem remains that the diverse factors, which influence disease progression are largely unknown, while tools for diagnosis have improved substantially.

We will identify patients for participation in a long-term clinical follow up study. Biomaterial (CSF, blood) will be obtained at baseline and subjected to a detailed protein analysis. In a subset of patients, a lumbar puncture will be repeated to compare baseline and follow up CSF. Within this study, a panel of proteins, comprising Aβ- and Tau-species as well as inflammation, glial and synaptic markers, potentially involved in disease progression will be measured in biomaterial from baseline and from follow up assessment. Clinical data will be correlated with the panel of disease and progression markers.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Alzheimer´s Disease

Exclusion Criteria:

Other neurological or psychiatric diseases Stroke

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients reporting to a memory clinic
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive Performance | 3-5 years
  performance in the ADAS cog test battery

SECONDARY OUTCOMES:
Biomarker | 3-5 years
  changes in the concentrations of biomarkers over time

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Peters, MD, Principal Investigator — Charité University Medicine, Psychiatry, CBF
Locations (1):
- Charité University Medicine, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No